CLINICAL TRIAL: NCT00967291
Title: Mitomycin and Ifosfamide (MI) as Salvage Therapy for Metastatic Pancreatic Adenocarcinoma: a Phase II Study.
Brief Title: Mitomycin C and Ifosfamide in Treating Patients With Metastatic Pancreatic Cancer
Acronym: PACT-11
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of activity and G3-4 toxicity at interim analysis
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Michele Reni, MD, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000642574; PACT-11 (Other: IRCCS San Raffaele); 2006-001163-29 (EudraCT Number)
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2009-08

CONDITIONS: Pancreatic Cancer
Keywords: acinar cell adenocarcinoma of the pancreas; duct cell adenocarcinoma of the pancreas; stage IV pancreatic cancer; recurrent pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Ifosfamide; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ifosfamide — 2,500 mg/mq on days 1-3 every 28 days
  Other Names: HOLOXAN
Drug: mitomycin C — 8 mg/mq on day 1 every 28 days
  Other Names: Mutamycin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as mitomycin C and ifosfamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving mitomycin C together with ifosfamide works in treating patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the therapeutic activity of a mitomycin C and ifosfamide combination, in terms of progression-free survival rate at 6 months, in patients with metastatic stage IV adenocarcinoma of the pancreas.

OUTLINE: Patients receive mitomycin C IV on day 1 and ifosfamide IV on days 1-3. Courses repeat every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas

  * Stage IV disease
  * Metastatic disease
* Prior treatment with gemcitabine-based chemotherapy, also in the adjuvant setting, with progression-free survival at ≤ 12 months
* Measurable disease according RECIST criteria
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100% (80-100% in patients > 70 years of age)
* Adequate bone marrow, liver, and kidney function
* Not pregnant or nursing
* No other prior or concurrent malignancies except surgically cured carcinoma in situ of the cervix, basal cell or squamous cell carcinoma of the skin, or other neoplasms with no evidence of disease ≥ 5 years
* No severe comorbidities that could compromise safety, including any of the following:

  * Cardiac failure
  * Cardiac arrhythmia
  * Prior myocardial infarction within the past 4 months
  * History of psychiatric disabilities

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior mitomycin C and ifosfamide
* No concurrent treatment with experimental drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Progression-free survival at 6 months | every 2 months during therapy; every 3 months thereafter
  CT scan

SECONDARY OUTCOMES:
Toxicity | monthly
  outpatient visit
Progression-free survival | every 2 months during therapy; every 3 months thereafter
  CT scan
Overall survival | monthly
  outpatient visit or phone interview

CONTACTS AND LOCATIONS:
Overall Officials: Michele Reni, MD, Principal Investigator — Istituto Scientifico H. San Raffaele
Locations (1):
- Istituto Scientifico H. San Raffaele, Milan, Italy